CLINICAL TRIAL: NCT01512628
Title: Hemostatic Changes After Colloid Fluid Administration During Total Hip Replacement Arthroplasty
Brief Title: Rotational Thromboelstometry (ROTEM) change_colloid_total Hip Replacement Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Assistant professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: B1111-140-010
Record Dates: First submitted 2012-01-09; First posted 2012-01-19 (Estimated); Last update posted 2014-01-28 (Estimated); Status verified 2014-01

CONDITIONS: Avascular Necrosis of Hip; Total Hip Replacement Arthroplasty
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- PENTA group (Active Comparator): Pentaspan is administered as a colloid.
  Interventions: Drug: Pentaspan, voluven, volulyte
- voluVEN group (Active Comparator): Voluven is administered as a colloid.
  Interventions: Drug: Pentaspan, voluven, volulyte
- voluLYTE group (Active Comparator): Volulyte is administered as a colloid.
  Interventions: Drug: Pentaspan, voluven, volulyte

INTERVENTIONS:
Drug: Pentaspan, voluven, volulyte — Different colloids are administered during operation for replacement of blood loss before the transfusion of blood.

SUMMARY:
The investigators administered different kinds of colloids before transfusion of red blood cell to patient undergoing total hip replacement arthroplasty. The investigators will compare the differences of changes in rotational thromboelastometry (ROTEM) data among them.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as avascular necrosis of hip and undergoing total hip replacement arthroplasty

Exclusion Criteria:

* hematologic disease
* anticoagulant medication
* preoperative hemoglobin < 10 g/dl
* renal disease
* pulmonary disease (pulmonary edema, effusion)
* cardiovascular disease (coronary heart disease, congestive heart failure)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2012-01; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
INTEM parameters change from preoperative values at post-operation | 30 minutes before operation and 30 minutes after operation
  clotting time (sec), clot firmness time (sec), alpah angle, maximum clot firmness (mm)
EXTEM parameters change from preoperative values at post-operation | 30 minutes before and 30 minutes after operation.
  clotting time (sec), clot firmness time (sec), alpah angle, maximum clot firmness (mm)
FIBTEM parameters change from preoperative values at post-operation | 30 min before and 30 min after operation
  maximum clot firmness (mm)

SECONDARY OUTCOMES:
Infused total fluid volume | Participants will be followed for the duration of THRA operation in operating room, an expected average tiem of 3 hours
  crystalloid and colloid
Hemoglobin | 30 minutes before operation and 30 minutes after operation
postoperative blood loss | postoperative 1 day and 2 day
Hematocrit | 30 minutes before operation and 30 minutes after operation
Platelet | 30 minutes before operation and 30 minutes after operation
Prothrombin Time-Internatiolnal Normalized Ratio | 30 minutes before operation and 30 minutes after operation
Activated Partial Thrombin Time | 30 minutes before operation and 30 minutes after operation
electrolytes | 30 minutes before operation and 30 minutes after operation

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam, Gyounggi, South Korea